CLINICAL TRIAL: NCT04153890
Title: Coaching End-of-Life Palliative Care for End-Stage Heart Failure Patients and Their Family Caregivers in Rural Appalachia
Brief Title: Family Palliative and End-of-Life Care for Advanced Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Ubolrat Piamjariyakul, Associate Dean for Research and Scholarship, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1709754988; 1R15NR018547-01 (NIH)
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure NYHA Class III; Heart Failure NYHA Class IV
Keywords: advanced heart failure, breathlessness, supportive care
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Intervention Model Description: This study is a low-risk randomized control trial design to test the implementation of the FamPALcare intervention with advanced HF patients and their primary family caregivers.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care provider and outcome assessor including data collectors will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FamPALcare (Experimental): FamPALcare: Intervention participants will receive standard care plus five weekly coaching sessions with telephone follow-up to reinforce HF palliative home care.
  Interventions: Behavioral: FamPALcare
- Standard Care (No Intervention): The standard care group will receive routine HF care and instruction at university hospital or at clinic.

INTERVENTIONS:
Behavioral: FamPALcare — Intervention participants will receive standard care plus five weekly coaching sessions with telephone follow-up to reinforce HF palliative home care.
  Arms: FamPALcare

SUMMARY:
Overall objective is to test whether the 5-weekly family home palliative and end-of-life care (FamPALcare) intervention educational and supportive sessions will improve rural home end-of-life and palliative care (EOLPC) for advanced heart failure at 6 months follow up.

DETAILED DESCRIPTION:
Heart failure (HF) afflicts 6.5 million Americans with devastating consequences to patients and their family caregivers especially during severe symptoms in the long-lasting end stage. Advanced HF was defined by American Heart Association (AHA) as "the presence of progressive and/or persistent severe signs and symptoms of HF despite optimized medical, surgical, and device therapy." When patients and family members are not prepared for worsening HF and are not informed about end-of-life and palliative care (EOLPC) conservative comfort options, they experience depression, fear of painful death, home care burden, and medical expenses from anxiously seeking aggressive but futile care. Notably, West Virginia (WV) has the highest HF death in the U.S. at 32.6 per 100,000 population, where 14% of those over 65 years have HF. WV is in the large Appalachian region, which stretches across eastern North America with 25.6 million people and contains a vast number of disadvantaged rural communities. National Institutes of Health has designated Appalachia as a high priority for research as residents experience extreme health and poverty inequities and limited access to healthcare. Furthermore, home EOLPC is lacking across this disadvantaged rural area. Thus, there is a need to investigate the new family intervention (FamPALcare), where nurses coach family-managed advanced HF care at home in Appalachia.

This study addresses the National Institutes of Health Academic Research Enhancement Award (AREA) priorities for conducting a low risk clinical trials to provide a foundation to advance scientific EOLPC knowledge and testing of our intervention efficacy in larger clinical trials. Additionally, effective EOLPC interventions are priorities of palliative care professionals and palliative care needs must be addressed with vulnerable and advanced HF patients and their families. This study also addresses the priority problem of the lack information for families providing advanced HF home care and preventing unwanted and unwarranted rehospitalizations at the advanced stage of HF.

This study uses a randomized controlled trial (RCT) design stratified by gender (male vs female) to determine any differences in the FamPALcare HF patients and their family caregiver outcomes versus standard care control group outcomes (N=72). Specific aims are to: (1) Test the FamPALcare nursing care intervention with patients and family members managing home supportive EOLPC for advanced HF in rural WV using a small randomized controlled trial (RCT) and (2) Assess implementation of the FamPALcare intervention and research procedures for subsequent clinical trials.

The control patients receive standard care given through the West Virginia University hospital and outpatient clinics, prescribed by the patient's cardiologist. The FamPALcare intervention group will receive standard care, plus 5-weekly FamPALcare intervention delivered by community-based nurses. FamPALcare intervention involves coaching patients and family caregivers in advanced HF home care and supporting EOLPC discussions. Data will be collected from all patients and caregivers independently at baseline, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Alert and consent to participate
2. Able to read and understand English
3. Advanced HF (NYHA III or IV), diagnosed by physician

Exclusion Criteria:

1. Already received or are on a waiting list for a heart transplant or left ventricular assist device (LVAD)
2. Diagnosed with a terminal illness or dementia, such as Alzheimer's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ubolrat Piamjariyakul, PhD, RN, Principal Investigator — West Virginia University, School of Nursing
Locations (1):
- West Virginia University Hospital, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The study plans to share data in aggregate and as overall study results.

REFERENCES:
- [Background] Piamjariyakul U, Petitte T, Smothers A, Wen S, Morrissey E, Young S, Sokos G, Moss AH, Smith CE. Study protocol of coaching end-of-life palliative care for advanced heart failure patients and their family caregivers in rural appalachia: a randomized controlled trial. BMC Palliat Care. 2019 Dec 29;18(1):119. doi: 10.1186/s12904-019-0500-z. PMID 31884945
- [Background] Piamjariyakul U, Keener TA, Smothers A, Young S, Shafique S, McDill S, Keech K, Petitte T, Pacheco C. Mentoring Undergraduate Nursing Students in Palliative Home Care Research. Teach Learn Nurs. 2021 Oct;16(4):423-428. doi: 10.1016/j.teln.2021.05.001. Epub 2021 Jun 5. No abstract available. PMID 34720774
- [Background] Piamjariyakul U, Shafique S, Friend DL, Adams KA, Sanghuachang W, Petitte TM, Young S. The development and evaluation of a short-term international student research and educational program. Int J Nurs Sci. 2023 Dec 6;11(1):83-90. doi: 10.1016/j.ijnss.2023.12.001. eCollection 2024 Jan. PMID 38352285
- [Result] Piamjariyakul U, Smothers A, Wang K, Shafique S, Wen S, Petitte T, Young S, Sokos G, Smith CE. Palliative care for patients with heart failure and family caregivers in rural Appalachia: a randomized controlled trial. BMC Palliat Care. 2024 Aug 3;23(1):199. doi: 10.1186/s12904-024-01531-2. PMID 39097733

RESULTS

PARTICIPANT FLOW:
Groups:
- FamPALcare- Patients; FamPALcare- Caregivers: Standard Care plus FamPALcare
  FamPALcare: Intervention participants will receive standard care plus five weekly coaching sessions with telephone follow-up to reinforce HF palliative home care.
- Standard Care- Patients; Standard Care- Caregivers: The standard care group will receive routine HF care and instruction at university hospital or at clinic appointments.
Period: Overall Study
Arm/Group | FamPALcare- Patients | Standard Care- Patients | FamPALcare- Caregivers | Standard Care- Caregivers
Started | 21 | 18 | 21 | 18
Completed | 12 | 16 | 12 | 16
Not Completed | 9 | 2 | 9 | 2
Not completed — Lost to Follow-up | 9 | 0 | 9 | 0
Not completed — Death | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FamPALcare- Patients | Standard Care- Patients | FamPALcare- Caregivers | Standard Care- Caregivers | Total
Number analyzed (Participants) | 21 | 18 | 21 | 18 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.57 (13.38) | 65.78 (14.51) | 64.19 (11.73) | 59.55 (14.57) | 63.86 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 16 | 14 | 43
  Male | 15 | 11 | 5 | 4 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 2 | 7
  White | 19 | 15 | 19 | 15 | 68
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 18 | 21 | 17 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 18 | 21 | 18 | 78

OUTCOME MEASURES:

1. Primary Outcome: Patient Heart Failure Health Status (KCCQ)- Baseline
Description: The patients Heart Failure Health Status was measured by administering the Kansas City Cardiomyopathy Questionnaire (KCCQ). KCCQ is a 12-item Likert scale (range 0-4). Total scores are calculated in a range of 0-100, with the higher score indicating better Heart Failure Health Status.
Time Frame: Baseline
Population: The overall number of participants will remain the same throughout the study timepoints as the data analysis was performed with the Intent-To-Treat (ITT) principle.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- FamPALcare: Standard Care plus FamPALcare
  FamPALcare: Intervention participants will receive standard care plus five weekly coaching sessions with telephone follow-up to reinforce HF palliative home care.
- Standard Care: The standard care group will receive routine HF care and instruction at university hospital or at clinic appointments.
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 26.79 (18.30) | 27.11 (14.63)

2. Primary Outcome: Patient Heart Failure Health Status (KCCQ) -3 Month
Description: as for outcome 1
Time Frame: 3 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 54.73 (22.58) | 44.57 (24.54)

3. Primary Outcome: Patient Heart Failure Health Status (KCCQ)- 6 Month
Description: as for outcome 1
Time Frame: 6 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 59.49 (21.29) | 46.00 (23.08)

4. Primary Outcome: Patient Mental Health - Patient Health Questionnaire (PHQ-4)- Baseline
Description: Patient-reported mental health measured by Patient Health Questionnaire (PHQ-4) of 4 questions. Each question is scored on a scale from 0 to 3, based on how often the respondent has been bothered by the problem 0 is not at all and 3 is nearly every day. The total score ranges from 0 to 12. The higher the score indicates a worse mental health status.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 5.71 (4.75) | 5.89 (3.67)

5. Primary Outcome: Patient Mental Health - Patient Health Questionnaire (PHQ4)- 3 Month
Description: as for outcome 4
Time Frame: 3 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 2.97 (2.46) | 3.90 (2.86)

6. Primary Outcome: Patient Mental Health - Patient Health Questionnaire (PHQ-4)- 6 Month
Description: as for outcome 4
Time Frame: 6 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Standard Care: The standard care group will receive routine HF care and instruction at university hospital or at clinic appointments. All patients can be referred for supportive care and heart failure care per national HF guidelines.
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 2.44 (1.89) | 4.10 (3.08)

7. Primary Outcome: Caregiver Mental Health - Patient Health Questionnaire (PHQ-4)- Baseline
Description: Caregiver mental health measured by Patient Health Questionnaire (PHQ-4) of 4 questions. Each question is scored on a scale from 0 to 3, based on how often the respondent has been bothered by the problem 0 is not at all and 3 is nearly every day. The total score ranges from 0 to 12. The higher the score indicates a worse mental health status.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 3.52 (3.72) | 4.33 (3.60)

8. Primary Outcome: Caregiver Mental Health - Patient Health Questionnaire (PHQ-4)- 3 Month
Description: as for outcome 7
Time Frame: 3 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 2.06 (1.64) | 4.53 (3.64)

9. Primary Outcome: Caregiver Mental Health - Patient Health Questionnaire (PHQ-4)- 6 Month
Description: as for outcome 7
Time Frame: 6 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 2.69 (2.01) | 4.32 (3.80)

10. Primary Outcome: Caregiver Quality of Life - SF12V2 Health Survey- Baseline (MCS-12)
Description: The SF-12v2 Health Survey is a multipurpose short-form questionnaire with only 12 questions with two summary scores, the SF-12 Physical Component Summary (PCS-12) and the SF-12 Mental Component Summary (MCS-12). The scoring range for the PCS-12 and MCS-12 is 0 to 100, with a lower score indicating a poorer level of Caregiver quality of life.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 45.85 (12.83) | 43.59 (11.91)

11. Primary Outcome: Caregiver Quality of Life - SF12v2 Health Survey- 3 Month (MCS-12)
Description: as for outcome 10
Time Frame: 3 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 47.55 (12.42) | 42.32 (17.08)

12. Primary Outcome: Caregiver Quality of Life - SF12v2 Health Survey- 6 Month (MCS-12)
Description: The SF-12v2 Health Survey is a multipurpose short-form questionnaire with only 12 questions with two summary scores, the SF-12 Physical Component Summary (PCS-12) and the SF-12 Mental Component Summary (MCS-12). The scoring range for both the PCS-12 and MCS-12 is 0 to 100, with a lower score indicating a poorer level of Caregiver quality of life.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 47.81 (13.44) | 46.32 (12.06)

13. Primary Outcome: Caregiver Quality of Life - SF12V2 Health Survey- Baseline (PCS-12)
Description: as for outcome 10
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 42.40 (13.99) | 40.48 (14.64)

14. Primary Outcome: Caregiver Quality of Life - SF12v2 Health Survey- 3 Month (PCS-12)
Description: as for outcome 10
Time Frame: 3 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 48.98 (11.07) | 40.66 (14.16)

15. Primary Outcome: Caregiver Quality of Life - SF12v2 Health Survey- 6 Month (PCS-12)
Description: as for outcome 10
Time Frame: 6 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 44.44 (16.35) | 41.87 (12.07)

16. Primary Outcome: Caregiver Burden (ZBI-12)- Baseline
Description: The Zarit Burden Interview-12 (ZBI-12) consists of 12 items that measure the emotional, physical, and social impact of caregiving. There are 12 questions and each question is rated on a 5-point scale from 0 (never) to 4 (nearly always). The total score ranges from 0 to 48, with higher scores indicating greater caregiver burden.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 8.12 (7.75) | 13.56 (9.76)

17. Primary Outcome: Caregiver Burden (ZBI-12)- 3 Month
Description: as for outcome 16
Time Frame: 3 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 9.48 (4.23) | 13.38 (7.02)

18. Primary Outcome: Caregiver Burden (ZBI-12)- 6 Month
Description: as for outcome 16
Time Frame: 6 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare | Standard Care
Number analyzed (Participants) | 21 | 18
score on a scale | 8.12 (3.67) | 9.93 (7.16)

19. Secondary Outcome: FamPALcare Helpfulness Scale
Description: This scale was completed voluntarily by participants that received the intervention (ARM Title: FamPALcare. The FamPALcare helpfulness scale is an 11-item Likert-type scale used to measure the perceived helpfulness of the FamPALcare intervention. Participants rate each item on a scale from 1 (not helpful) to 5 (very helpful). This scale is used to assess the effectiveness of the intervention in improving outcomes for patients with heart failure and their caregivers.
Time Frame: 6 months
Population: This was a voluntary questionnaire by participants that had received the intervention. All intervention participants (patients and caregivers) that completed the study were provided with this survey. The number pf participants analyzed represents those that completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FamPALcare
Number analyzed (Participants) | 9
score on a scale | 4.46 (0.49)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse Event information was collected during the follow up care visits in both the intervention arm and the standard care arm.
Arm/Group | FamPALcare- Patients | Standard Care- Patients | FamPALcare- Caregivers | Standard Care- Caregivers
All-Cause Mortality (participants affected / at risk) | 0/21 | 2/18 | 0/21 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/18 | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 0/21 | 0/18 | 0/21 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FamPALcare- Patients (N=21) | Standard Care- Patients (N=18) | FamPALcare- Caregivers (N=21) | Standard Care- Caregivers (N=18)
Death (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
There was an expected delay in our initial enrollment during winter (December to March) due to extreme weather and road conditions in rural Appalachia and COVID-19 restrictions (December 2019 through Mid-2022). However, only slight variation in participant intervention timelines was necessary in a few cases. The flexibility of the intervention schedule helped with the retention of participants in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT04153890/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT04153890/ICF_001.pdf